CLINICAL TRIAL: NCT02271620
Title: The Prevalence and Clinical Characteristics of Children With Local Allergic Rhinitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Orathai Piboonpocanun, Division of allergy and immunology, Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 759/25569(EC3)
Record Dates: First submitted 2014-09-09; First posted 2014-10-22 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Other Allergic Rhinitis
Keywords: 1 prevalence; 2 children; 3 local allergic rhinitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- nonallergic rhinitis (Other): nonallergic rhinitis nasal allergen provocation test
  Interventions: Procedure: nasal allergen provocation test

INTERVENTIONS:
Procedure: nasal allergen provocation test — nasal allergen provocation test

SUMMARY:
* To determine prevalence of local allergic rhinitis (LAR)
* To evaluate clinical characteristic and severity of local allergic rhinitis
* To measure changing of tryptase and Specific IgE for Dermatophagoides pteronyssinus (Dp) after nasal allergen provocation test (NAPT)

DETAILED DESCRIPTION:
Children 8-18 years with NAR were recruited. A NAPT with Der p 1 solutions (NAPT-DP) at 200 AU/mL, 600 AU/mL and 2000 AU/mL at 15-minute interval was performed, respectively. The immediate responses to NAPT-DP were assessed using symptoms score, peak nasal inspiratory flow (PNIF) and acoustic rhinometry (ARM). The nasal tryptase and sIgE-DP were measured at baseline, 15 min and 1 h after positive NAPT-DP. Allergic rhinitis (AR) patients were used as positive control.

ELIGIBILITY:
Inclusion Criteria:

* Children 8-15 years who were diagnosed with nonallergic rhinitis (NAR) at least 1 year
* No respiratory infections in the previous 4 weeks
* No following treatment of
* systemic corticosteroid 4 weeks
* intranasal corticosteroid 2 weeks
* oral antihistamine 1 week
* leukotriene antagonist 1 week

Exclusion Criteria:

* Patients with underlying disease:
* chronic rhinosinusitis and nasal polyp
* immunological disease
* chronic renal disease
* hepatobiliary disease
* cardiovascular disease
* cancer
* Parental withdraw consent
* Patient with uncontrolled asthma, peak expiratory flow rate (PEFR) < 80% of predicted

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
prevalence of local allergic rhinitis (LAR) | 1 year
  positive nasal allergen provocation test with Der p1

CONTACTS AND LOCATIONS:
Overall Officials: Orathai Piboonpocanun, assoc. prof., Principal Investigator — 66815818803
Locations (2):
- Thailand (2):
  - Division of allergy and immunology, Department of pediatric, Siriraj Hospital, Bangkoknoi, Bangkok
  - Division of Allergy and Immunology, Department of Pediatrics, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok

IPD SHARING:
Plan to Share IPD: No